CLINICAL TRIAL: NCT02924233
Title: An Open-label, Randomized, Multicenter, Phase 1b/2b Trial Investigating the Safety and Preliminary Antitumor Effects of Sym004 in Combination With Nivolumab Versus Nivolumab Monotherapy in EGFR-amplified Squamous Non-Small Cell Lung Cancer
Brief Title: Sym004 in Combination With Nivolumab Versus Nivolumab Monotherapy in EGFR-amplified Squamous Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Symphogen made a business decision to no longer perform the clinical study
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-10
Record Dates: First submitted 2016-09-28; First posted 2016-10-05 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Squamous Non-Small Cell Lung Cancer
Keywords: Squamous; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — futuximab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sym004 + nivolumab (Experimental): Phase 1b, dose-escalation:
  Dose Level 1: Sym004 + nivolumab (Q2W)
  Dose Level 2: Sym004 + nivolumab (Q2W)
  Dose Level -1: Sym004 + nivolumab, if needed
  Interventions: Drug: Sym004; Drug: Nivolumab
- Sym004 (RP2D) + nivolumab (Experimental): Phase 2b, dose-expansion:
  Receiving Sym004 in the RP2D in combination with nivolumab (Q2W)
  Interventions: Drug: Sym004; Drug: Nivolumab
- Nivolumab (Active Comparator): Phase 2b, dose-expansion:
  Receiving nivolumab monotherapy (Q2W)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Sym004 — Sym004 is a 1:1 mixture of two monoclonal antibodies (mAbs) which bind to two non-overlapping epitopes of the Epidermal Growth Factor Receptor (EGFR).
  Sym004 will be administered at different dose-levels via infusion Q2W
  Arms: Sym004 (RP2D) + nivolumab; Sym004 + nivolumab
Drug: Nivolumab — Nivolumab is a humanized immunoglobulin G4 (IgG4) anti-PD-1 monoclonal antibody. Nivolumab will be administered via 60-minute infusion Q2W

SUMMARY:
This is a phase 1b/2b study investigating the safety and preliminary antitumor effects of Sym004 in combination with nivolumab versus nivolumab monotherapy when administered every second week.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated written informed consent
* Male or female ≥18 years of age at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy >3 months assessed during Screening
* Histologically or cytologically confirmed, locally advanced or metastatic squamous NSCLC

Main Exclusion Criteria:

* Any antineoplastic agent (standard or investigational) within 2 weeks prior to starting trial treatment
* Radiosurgery or radiotherapy for target lesions within 2 weeks prior to starting trial treatment
* Prophylactic use of hematopoietic growth factors within 1 week prior to starting trial treatment
* Active Central Nervous System (CNS) metastases or carcinomatous meningitis
* Women who are pregnant
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Determination of the Dose-Limiting Toxicities (DLT) and the MTD and/or RP2D of escalating doses of Sym004 in combination with a standard dose of nivolumab | 1 year
Phase 2b: Evaluation of the antitumor effects of the RP2D of Sym004 when administered in combination with a standard dose of nivolumab as measured by Response Rate | 1.5 years

IPD SHARING:
Plan to Share IPD: Undecided